CLINICAL TRIAL: NCT02147587
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Study To Assess The Immune Response Following Administration Of Zoster Vaccine To Subjects With Rheumatoid Arthritis Receiving Tofacitinib (Cp-690,550) Or Placebo With Background Methotrexate Treatment
Brief Title: A Study to Assess Immune Response Following Zoster Vaccination to Subjects With Rheumatoid Arthritis Receiving Tofacitinib or Placebo With Background Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3921237; 2014-000706-34 (EudraCT Number)
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Results first posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tofacitinib 5 mg BID (oral) (70 subjects) (Experimental): Zoster vaccine will be administered to subjects on background methotrexate; treatment with 5 mg tofacitinib twice daily will begin 2 to 3 weeks following vaccination and continue for 12 weeks.
  Interventions: Drug: Tofacitinib
- Placebo tofacitinib BID (oral) (70 subjects) (Placebo Comparator): Zoster vaccine will be administered to subjects on background methotrexate; treatment with placebo twice daily will begin 2 to 3 weeks following vaccination and continue for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tofacitinib — 5 mg twice daily of tofacitinib with background methotrexate for 12 weeks
  Arms: Tofacitinib 5 mg BID (oral) (70 subjects)
Drug: Placebo — Placebo tablets twice daily with background methotrexate for 12 weeks
  Arms: Placebo tofacitinib BID (oral) (70 subjects)

SUMMARY:
This study will evaluate immune response following administration of zoster vaccine in subjects with rheumatoid arthritis who are receiving background methotrexate and initiate 5 mg twice daily of tofacitinib or placebo for tofacitinib 2 to 3 weeks following vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have moderate to severe rheumatoid arthritis inadequately controlled by methotrexate as defined by the American College of Rheumatology (ACR) classification criteria for Rheumatoid arthritis, painful and swollen joint counts and C-reactive protein (CRP).
* Screening CRP >3 mg/L or CDAI score > 10 at screening or at baseline before vaccination.
* Subjects must have active disease at screening and baseline.
* Must be at least 50 years of age or older.

Exclusion Criteria:

* History of receiving any varicella-zoster virus vaccine
* Receipt of any vaccines within 6 weeks of first dose of study treatment.
* Subjects with current infections or history of infections.
* History of recurrent (more than one episode) of herpes zoster or disseminated (a single episode) of herpes zoster or disseminated (a single episode) of herpes simplex.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (36):
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Drug Shipping Address (IRB# 14-000826) Ronald Regan, Los Angeles, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Center for Arthritis and Rheumatic Diseases, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - Florida Arthritis and Osteoporosis Center, Port Richey, Florida
  - Gulf Coast Medical Center, Port Richey, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Suncoast Medical Clinic, St. Petersburg, Florida
  - Sun Coast Medical Clinic, St. Petersburg, Florida
  - Health Point Medical Group, Inc., Tampa, Florida
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Diagnostic Rheumatology And Research, PC, Indianapolis, Indiana
  - Arthritis Treatment Center, Frederick, Maryland
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The Center for Rheumatology, LLP, Albany, New York
  - Buffalo Rheumatology and Medicine, PLLC, Orchard Park, New York
  - Piedmont Rheumatology, P.A, Hickory, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Novant Health Imaging Julian Road, Salisbury, North Carolina
  - East Penn Rheumatology Associates, PC, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading LLP, Wyomissing, Pennsylvania
  - Palmetto Clinical Trial Services, LLC, Greenville, South Carolina
  - Arthritis Clinic, Jackson, Tennessee
  - West Tennessee Research Institute, Jackson, Tennessee
  - Rheumatology Consultants, PLLC, Knoxville, Tennessee
  - Office of John P. Lavery, MD, PA, Allen, Texas
  - Baylor Research Institute Arthritis Care and Research Center, Dallas, Texas
  - The Vancouver Clinic (Drug Shipment Only), Vancouver, Washington
  - The Vancouver Clinic, Inc, PS, Vancouver, Washington

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Winthrop KL, Wouters AG, Choy EH, Soma K, Hodge JA, Nduaka CI, Biswas P, Needle E, Passador S, Mojcik CF, Rigby WF. The Safety and Immunogenicity of Live Zoster Vaccination in Patients With Rheumatoid Arthritis Before Starting Tofacitinib: A Randomized Phase II Trial. Arthritis Rheumatol. 2017 Oct;69(10):1969-1977. doi: 10.1002/art.40187. Epub 2017 Sep 6. PMID 28845577
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921237&StudyName=A%20Study%20to%20Assess%20Immune%20Response%20Following%20Zoster%20Vaccination%20to%20Subjects%20with%20Rheumatoid%20Arthritis%20Receiving%20Tofacitinib%20or%20Placebo%20with

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The zoster vaccine was administered at least 2 weeks (14 to 21 days) prior to initiation of CP-690,550 (tofacitinib) or placebo in rheumatoid arthritis (RA) participants on background methotrexate therapy.
Groups:
- Placebo Twice a Day: Following administration of zoster vaccine, participants with Rheumatoid Arthritis (RA) on background methotrexate received placebo matched tofacitinib tablets twice a day orally for up to 12 weeks.
- Tofacitinib 5 mg Twice a Day: Following administration of zoster vaccine to RA participants receiving background methotrexate, participants received tofacitinib 5 mg twice a day orally for up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo Twice a Day | Tofacitinib 5 mg Twice a Day
Started | 57 | 55
Completed | 46 | 50
Not Completed | 11 | 5
Not completed — Adverse Event | 9 | 4
Not completed — Lack of Efficacy | 2 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all randomized participants who received at least 1 dose of study drug (tofacitinib or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Twice a Day | Tofacitinib 5 mg Twice a Day | Total
Number analyzed (Participants) | 57 | 55 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (8.7) | 61.7 (6.2) | 61.8 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 42 | 80
  Male | 19 | 13 | 32

OUTCOME MEASURES:

1. Primary Outcome: Fold Change From Baseline in Varicella Zoster Virus (VZV)-Specific Immunoglobulin G (IgG) Levels at Week 4
Description: VZV-specific IgG levels as measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline (pre-vaccination; Day -14), Week 4 (6 weeks post-vaccination)
Population: The evaluable immunogenicity analysis population included randomized participants who had at least 1 dose of study drug (tofacitinib or placebo) and who complied closely with protocol eligibility criteria, visit windows for study procedures, had valid assay results at the primary visits and no major protocol deviations.
Measure: Geometric Mean (80% Confidence Interval); unit: fold rise
Arm/Group | Placebo Twice a Day | Tofacitinib 5 mg Twice a Day
Number analyzed (Participants) | 53 | 54
fold rise | 1.736 [1.546 to 1.950] | 2.105 [1.871 to 2.369]
Statistical Analysis 1: Comparison: Placebo Twice a Day vs Tofacitinib 5 mg Twice a Day; Geometric Mean Fold Rise (GMFR) for Tofacitinib versus Placebo (Week 4); Test type: Superiority or Other; ANCOVA; Repeated-measures ANCOVA model for the log-transformed GMFRs are adjusted for baseline factors. GMFRs and 80% CIs are back-transformed from log scale; Ratio of GMFR = 1.213, 80% CI 2-sided [1.033 to 1.424] — Ratio of GMFRs (Tofacitinib/Placebo) at Week 4

2. Secondary Outcome: Fold Change From Baseline in VZV-Specific IgG Levels at Day 1 and Week 12
Time Frame: Baseline (pre-vaccination; Day -14), Day 1 (2 weeks post-vaccination), Week 12 (14 weeks post-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (80% Confidence Interval); unit: fold rise
Arm/Group | Placebo Twice a Day | Tofacitinib 5 mg Twice a Day
Number analyzed (Participants) | 53 | 54
fold rise
  Day 1 | 1.947 [1.733 to 2.186] | 2.005 [1.782 to 2.256]
  Week 12: number analyzed (Participants) | 44 | 48
  Week 12 | 1.496 [1.323 to 1.691] | 1.636 [1.448 to 1.847]
Statistical Analysis 1: Comparison: Placebo Twice a Day vs Tofacitinib 5 mg Twice a Day; GMFR for Tofacitinib versus Placebo (Day 1); Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of GMFR = 1.030, 80% CI 2-sided [0.877 to 1.209] — Ratio of GMFRs (Tofacitinib/Placebo) at Day 1
Statistical Analysis 2: Comparison: Placebo Twice a Day vs Tofacitinib 5 mg Twice a Day; GMFR for Tofacitinib versus Placebo (Week 12); Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of GMFR = 1.093, 80% CI 2-sided [0.924 to 1.294] — Ratio of GMFRs (Tofacitinib/Placebo) at Week 12

3. Secondary Outcome: Absolute Values in VZV-Specific IgG Levels at Day 1, Week 4 and Week 12
Description: The absolute geometric mean titer (GMT) of VZV-specific IgG levels was calculated from logarithmically transformed assay values.
Time Frame: Day 1 (2 weeks post-vaccination), Week 4 (6 weeks post-vaccination), Week 12 (14 weeks post-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (80% Confidence Interval); unit: [gp]ELISA units/mL
Arm/Group | Placebo Twice a Day | Tofacitinib 5 mg Twice a Day
Number analyzed (Participants) | 53 | 54
[gp]ELISA units/mL
  Day 1 | 361.603 [300.012 to 435.838] | 384.219 [317.477 to 464.993]
  Week 4 | 322.486 [267.557 to 388.690] | 403.422 [333.343 to 488.232]
  Week 12: number analyzed (Participants) | 44 | 48
  Week 12 | 278.599 [229.984 to 337.489] | 312.328 [257.319 to 379.096]
Statistical Analysis 1: Comparison: Placebo Twice a Day vs Tofacitinib 5 mg Twice a Day; Geometric Mean Titer (GMT) for Tofacitinib versus Placebo (Day 1); Test type: Superiority or Other; ANCOVA; Repeated-measures ANCOVA model for the log-transformed GMTs are adjusted for baseline factors. GMTs and 80% CIs are back-transformed from log scale; Ratio of GMT = 1.063, 80% CI 2-sided [0.821 to 1.375] — Ratio of GMTs (Tofacitinib/Placebo) at Day 1
Statistical Analysis 2: Comparison: Placebo Twice a Day vs Tofacitinib 5 mg Twice a Day; GMT for Tofacitinib versus Placebo (Week 4); Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 3, analysis 1]; Ratio of GMT = 1.251, 80% CI 2-sided [0.967 to 1.618] — Ratio of GMTs (Tofacitinib/Placebo) at Week 4
Statistical Analysis 3: Comparison: Placebo Twice a Day vs Tofacitinib 5 mg Twice a Day; GMT for Tofacitinib versus Placebo (Week 12); Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 3, analysis 1]; Ratio of GMT = 1.121, 80% CI 2-sided [0.862 to 1.459] — Ratio of GMTs (Tofacitinib/Placebo) at Week 12

4. Secondary Outcome: Percentage of Participants With >=1.5 Fold Change in VZV-Specific IgG Levels Day 1, Week 4 and Week 12
Description: VZV-specific IgG levels as measured by ELISA. A ratio greater than or equal to (>=)1.5 was defined as a responder.
Time Frame: Day 1 (2 weeks post-vaccination), Week 4 (6 weeks post-vaccination), Week 12 (14 weeks post-vaccination)
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Twice a Day | Tofacitinib 5 mg Twice a Day
Number analyzed (Participants) | 53 | 54
percentage of participants
  Day 1 | 47.17 [37.66 to 56.85] | 55.56 [45.93 to 64.86]
  Week 4 | 43.40 [34.06 to 53.13] | 57.41 [47.77 to 66.61]
  Week 12: number analyzed (Participants) | 44 | 48
  Week 12 | 43.18 [32.90 to 53.96] | 45.83 [35.87 to 56.07]
Statistical Analysis 1: Comparison: Placebo Twice a Day vs Tofacitinib 5 mg Twice a Day; Tofacitinib versus Placebo (Day 1); Test type: Superiority or Other; 80% CI based on Chan and Zhang method; Difference in percentages = 8.39, 80% CI 2-sided [-4.05 to 20.56]
Statistical Analysis 2: Comparison: Placebo Twice a Day vs Tofacitinib 5 mg Twice a Day; Tofacitinib versus Placebo (Week 4); Test type: Superiority or Other; 80% CI based on Chan and Zhang method; Difference in percentages = 14.01, 80% CI 2-sided [1.57 to 26.03]
Statistical Analysis 3: Comparison: Placebo Twice a Day vs Tofacitinib 5 mg Twice a Day; Tofacitinib versus Placebo (Week 12); Test type: Superiority or Other; 80% CI based on Chan and Zhang method; Difference in percentages = 2.65, 80% CI 2-sided [-10.66 to 15.83]

5. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 16 that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to Week 16
Population: The safety analysis population included randomized participants who received at least 1 dose of the study drug (tofacitinib or placebo).
Measure: Number; unit: participants
Arm/Group | Placebo Twice a Day | Tofacitinib 5 mg Twice a Day
Number analyzed (Participants) | 57 | 55
participants
  AEs | 21 | 16
  SAEs | 0 | 3

6. Other Pre Specified Outcome: Number of Participants With Zoster Vaccine-Related AEs by System Organ Class
Description: Zoster vaccine-related AEs included General Disorders and Administration Site Conditions (injection site erythema, pain, pruritis, rash, swelling; vaccination site erythema, pruritus, rash), Infections and Infestations (disseminated herpes zoster), and Musculoskeletal and Connective Tissue Disorders (myalgia). All zoster vaccine-related AEs were mild, except for the herpes zoster AE classified under Infections and Infestations, which was moderate in severity.
Time Frame: Baseline up to Week 16
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo Twice a Day | Tofacitinib 5 mg Twice a Day
Number analyzed (Participants) | 57 | 55
participants
  General and Administration Site Conditions | 2 | 4
  Infections and Infestations | 0 | 1
  Musculoskeletal and Connective Tissue Disorders | 0 | 1

7. Other Pre Specified Outcome: Number of Participants With Clinical Herpes Zoster Events by Severity
Description: Clinical herpes is manifested as mild, moderate, or severe disseminated herpes zoster.
Time Frame: Baseline up to Week 16
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo Twice a Day | Tofacitinib 5 mg Twice a Day
Number analyzed (Participants) | 57 | 55
participants
  Mild Herpes Zoster | 0 | 0
  Moderate Herpes Zoster | 0 | 1
  Severe Herpes Zoster | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Parameters
Description: Participants with the following abnormalities were discontinued from the study: 2 sequential absolute neutrophil counts (ANC) <1000/mm^3; 2 sequential hemoglobin values <8.0 g/dL or decreases of >30% from baseline value; 2 sequential absolute lymphocyte count <500/mm^3; 2 sequential platelet counts <75,000/mm^3; 2 sequential alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevations >=3 times the upper limit of normal (X ULN) with a total bilirubin value >=2X ULN, elevated international normalized ratio (INR), or accompanied by signs/symptoms consistent with hepatic injury; 2 sequential ALT or AST elevations >=5X ULN regardless of total bilirubin or accompanying symptoms; confirmed increases in serum creatinine (SCr) >50% over the average of screening and baseline values; a confirmed positive urine pregnancy test or refusal to use appropriate contraception in a woman of childbearing potential.
Time Frame: Baseline up to Week 16
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo Twice a Day | Tofacitinib 5 mg Twice a Day
Number analyzed (Participants) | 57 | 55
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo Twice a Day | Tofacitinib 5 mg Twice a Day
Serious Adverse Events (participants affected / at risk) | 0/57 | 3/55
Other Adverse Events (participants affected / at risk) | 9/57 | 6/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Twice a Day (N=57) | Tofacitinib 5 mg Twice a Day (N=55)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) — Bile duct stone and cholangitis occurred in the same subject.
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Bile duct stone and cholangitis occurred in the same subject.
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 1 (1) — adjudicated AE term "vaccine dissemination VZV"
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Twice a Day (N=57) | Tofacitinib 5 mg Twice a Day (N=55)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.